CLINICAL TRIAL: NCT06280209
Title: A Phase 1/2, Open-Label, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Intravenous Doses of BMN 351 in Participants With Duchenne Muscular Dystrophy
Brief Title: A Phase 1/2 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMN 351 in Participants With Duchenne Muscular Dystrophy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 351-201; 2023-506737-30-00 (Other: EU CT)
Record Dates: First submitted 2024-01-26; First posted 2024-02-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1A (Experimental): Cohort 1A will consist of both a single ascending dose (SAD) part and a multiple ascending dose (MAD). BMN 351 will be administered once every 2 weeks during the SAD portion of the study for up to 8 weeks and once weekly during the MAD portion for up to 89 weeks.
  Interventions: Drug: BMN 351
- Cohort 1B (Experimental): BMN 351 low dose will be administered once weekly for up to 97 weeks
  Interventions: Drug: BMN 351
- Cohort 2 (Experimental): BMN 351 medium dose will be administered once weekly for up to 73 weeks
  Interventions: Drug: BMN 351
- Cohort 3 (Experimental): BMN 351 high dose will be administered once weekly for up to 48 weeks
  Interventions: Drug: BMN 351

INTERVENTIONS:
Drug: BMN 351 — Anti-sense Oligonucleotide BMN 351 will be administered intravenously.

SUMMARY:
The purpose of this study is to test the safety and tolerability of BMN 351 in participants with Duchenne Muscular Dystrophy (DMD) with a genetic mutation amenable to exon 51 skipping.

DETAILED DESCRIPTION:
This is Phase 1/2, open-label, multi-center study consisting of 2 parts to evaluate the safety and tolerability of BMN 351 at escalating doses in participants with Duchenne Muscular Dystrophy (DMD) with genetic mutations amenable to exon 51 skipping.

Participants will be assigned to one of three groups called cohorts (Cohort 1, 2 or 3). Cohort 1 participants are further divided into Cohort 1A and Cohort 1B. In Cohort 1A, 3 participants will receive increasing doses once every 2 weeks with a visit to assess safety measures collected the week after dosing prior to escalating doses of BMN 351. In part 2, the participants in cohort 1A will transition to once weekly dosing. The participants in Cohort 1B, 2, and 3 will initiate low, medium, and high doses of BMN 351 and continue once weekly dosing at that same dose. The study will enroll approximately 18 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 10
* Diagnosis of Duchenne muscular dystrophy with a specific genetic change amenable to exon 51 skipping
* Able to walk
* Not requiring assistance from a ventilator to breathe
* Currently on consistent doses of steroid treatment for the last 12 weeks

Exclusion Criteria:

* The participant will have some initial clinical labs and studies to assess baseline level of heart and lung function.
* Treatment with an exon skipping therapy within 12 weeks prior to the first visit.
* Any history of treatment with gene therapy

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate and safety and tolerability of single and multiple doses of BMN 351 (incidence, severity, and dose-relationship of adverse effects and changes in laboratory parameters). | Up to 97 weeks.
  The safety and tolerability of BMN 351 will be assessed based on the incidence of adverse and serious adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) concentration of BMN 351 in plasma, urine and muscle approximately every 8 weeks for up to 97 weeks. | Serial measurements pre and post infusion.
  Serial measurements of plasma and urine PK predose approximately hourly up to 24 hours post-infusion. Muscle PK will be measured at 13 weeks or 25 weeks only post dosing.

OTHER OUTCOMES:
To evaluate the immune response to BMN 351. | Up to 97 weeks
  Anti-BMN 351 antibodies, anti-dystrophin antibodies.
To evaluate the effect of BMN 351 on physical function. | Change from baseline at week 25.
  Change from baseline on 6 Minute Walk Test (6MWT).
To evaluate the effect of BMN 351 on physical function. | Change from baseline at week 25.
  Change from baseline on North Star Ambulatory Assessment (NSAA).
Change from baseline in dystrophin expression measured by Liquid chromatography-mass spectrometry (LC-MS). | Baseline, Week 13 or Week 25

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (2):
  - Fondazione Serena Onlus - Centro Clinico NeMO Milano, Milan
  - UOC Fase I - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Viamed Santa Angela De la Cruz, Seville
- Yeditepe University Kosuyolu Hospital, Istanbul, Turkey (Türkiye)
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom